CLINICAL TRIAL: NCT03418519
Title: A Comparative Analysis on Physical Activity Performance and Motor Function of Affected Upper Extremity Before and After a CIMT Program in Young Children With Hemiparetic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Yi Kwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-11-120
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Hemiplegic Cerebral Palsy With Spasticity (Diagnosis)
MeSH Terms: conditions — Disease | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIMT group (Experimental): Two-hour mCIMT per day for 15 days (dosage = 30 hours)
  24-hour restraint for 3 weeks
  Interventions: Other: Constraint Induced Movement Therapy
- Control group (No Intervention): no CIMT

INTERVENTIONS:
Other: Constraint Induced Movement Therapy — Constraint-induced movement therapy (CIMT) is a high-dosage, efficacious, rehabilitation approach used for children with hemiplegic cerebral palsy
  Other Names: CIMT
  Arms: CIMT group

SUMMARY:
This study evaluates CIMT(Constraint Induced Movement Therapy) in the treatment of physical activity performance and motor function of the weaker extremity in young children with cerebral palsy. Half of participants will receive CIMT while the other half will receive no treatment.

DETAILED DESCRIPTION:
Constraint-induced movement therapy (CIMT) is a short-term, intensive treatment to promote functional arm and hand skills in people with hemiparesis. It usually involves constraint of the non-involved extremity and intensive movement practice of the weaker extremity.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with spastic hemiplegic cerebral palsy
* age between 18 months and 36 months
* Mini-MACS level 1-4

Exclusion Criteria:

* botox injection in upper extremity within 6 months
* poor cooperation with cognitive impairment
* any musculoskeletal disease
* visual or hearing impairment
* uncontrollable epilepsy
* skin damage that makes impossible for participant to wear a splint
* Mini-MACS level 5

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2018-01-09 (Actual); Primary Completion 2019-04-08 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Accelerometers(physical activity performance) | 3 days
  For the upper limb use assessment, participants wear two accelerometers (one on each wrist). To quantify the affected upper limb movement relative to the unaffected upper limb before and after the CIMT program, two other variables are computed: use ratio and magnitude ratio. The use ratio is the ratio of the active duration for the affected arm to that for the unaffected arm. The magnitude ratio quantifies the contribution of the affected upper limb to activity.
Pediatric Motor Activity Log(PMAL) | 30 minutes
  The Pediatric Motor Activity Log (PMAL) is a parent-report measure of the use, by children with hemiplegic cerebral palsy, of their affected upper limb in everyday activities. Each item is scored 0-5(0= Never used affected arm , 5= Used affected arm on almost every occasion)

SECONDARY OUTCOMES:
Pediatric Evaluation of Disability Inventory(PEDI) | 30 minutes
  The PEDI is a parental-report, or structured-interview, instrument used by pediatric physical therapists and other rehabilitation professionals to assess functional abilities of young children children
Peabody Developmental Motor Scales-2(PDMS-2) | 30 minutes
  The PDMS-2 consists of six subtests: Reflexes (for children from birth through 11 months), Stationary (ability to sustain control of body within its center of gravity), Locomotion (ability to move from one place to another), Object Manipulation (ability to manipulate balls for children 12 months and older), Grasping (ability to use hands), and Visual-Motor Integration (ability to use visual perpetual skills to perform complex eye-hand coordination tasks).
Gross motor function measure - 66(GMFM-66) | 30 minutes
  The 88 items of the GMFM are measured by observation of the child and scored on a 4-point ordinal scale (0=does not initiate, 1=initiates <10% of activity, 2=partially completes 10% to <100% of activity, 3=completes activity). The items are weighted equally and grouped into 5 dimensions: (1) lying and rolling (17 items), (2) sitting (20 items), (3) crawling and kneeling (14 items), (4) standing (13 items), and (5) walking, running, jumping (24 items).

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Hwang YS, Kwon JY. Effects of Modified Constraint-Induced Movement Therapy in Real-World Arm Use in Young Children with Unilateral Cerebral Palsy: A Single-Blind Randomized Trial. Neuropediatrics. 2020 Aug;51(4):259-266. doi: 10.1055/s-0040-1702220. Epub 2020 Mar 6. PMID 32143221